CLINICAL TRIAL: NCT05172895
Title: Clinical Characteristics and Pathogenic Mechanisms of Anemia in Celiac Disease
Brief Title: Characteristics of Anemia in Celiac Disease
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, Principal Investigator, University of Palermo
Other Study IDs: ACPM28
Record Dates: First submitted 2021-11-30; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Prevalence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Presence, prevalence, severity, and morphological characteristics of anemia — Evaluation of the presence, prevalence, severity, and morphological characteristics of anemia, trying to define, when possible, the underlying pathogenetic mechanisms, paying particular attention to the characteristics of menstrual cycles, the iron, folate and vitamin B12 metabolism, any chronic inflammatory state, and thyroid hormones.
Other: Effect of gluten-free diet on anemia — Evaluation of the therapeutic responses (i.e., improvement/regression) of anemia after at least one year of GFD.

SUMMARY:
Celiac Disease (CD) is an autoimmune disease involving the mucosa of the small intestine, triggered by the ingestion of gluten in genetically predisposed individuals. CD represents a global health problem. The clinical presentation of CD is characterized by a broad spectrum of both intestinal and extraintestinal manifestations, involving one or more organs. Anemia is one of the most common extraintestinal clinical manifestations of CD, present in more than half of adult patients at the time of diagnosis. Anemia in CD has a multifactorial pathogenesis: a) lack of absorption (or, sometimes, loss, as in the case of iron), of some micronutrients, such as iron, folate, vitamin B12, copper and zinc, b) coexistence of a chronic inflammatory state, as in the case of inflammatory bowel disease (IBD), c) refractory CD, d) medullary aplasia. The main purpose of this multicentre research is to evaluate, retrospectively, analyzing the clinical and laboratory data of CD patients, the presence, prevalence, severity, and morphological characteristics of anemia, trying to define, when possible, the underlying pathogenetic mechanisms, paying particular attention to the characteristics of menstrual cycles, the iron, folate and vitamin B12 metabolism, any chronic inflammatory state, and thyroid hormones. It will be also recorded, in a subgroup of the selected CD patients, any therapeutic responses (i.e., improvement/regression) of anemia after at least one year of GFD.

DETAILED DESCRIPTION:
Celiac Disease (CD) is an autoimmune disease involving the mucosa of the small intestine, triggered by the ingestion of gluten in genetically predisposed individuals. CD represents a global health problem. The prevalence of CD, confirmed by intestinal biopsy, is estimated to be over 1% of the population of the Western world. Interestingly, the incidence of CD is continuously increasing around the world. CD is more common in women and children, although it is also becoming a common diagnosis also in men and adults. The clinical presentation of CD is characterized by a broad spectrum of both intestinal and extraintestinal manifestations, involving one or more organs. Several clinical categories of CD have been identified, including classical/typical CD (characterized by intestinal symptoms), atypical/subclinical CD (characterized by minor or extraintestinal symptoms), and silent CD (characterized by no symptoms). The category of "potential" CD was established for those patients with positive serology but without crypt hyperplasia and villous atrophy on duodenal biopsy. Duodenal biopsies can be avoided in the pediatric population, with high positive titer of IgA class anti-tTG (>10 times the upper limit of normal), associated with EMA-positivity. The treatment of CD is based on gluten-free diet (GFD).

Anemia is one of the most common extraintestinal clinical manifestations of CD, present in more than half of adult patients at the time of diagnosis. Anemia in CD has a multifactorial pathogenesis: a) lack of absorption (or, sometimes, loss, as in the case of iron), of some micronutrients, such as iron, folate, vitamin B12, copper and zinc, b) coexistence of a chronic inflammatory state, as in the case of inflammatory bowel disease (IBD), c) refractory CD, d) medullary aplasia.

The main purpose of this multicentre research is to evaluate, retrospectively, analyzing the clinical and laboratory data of CD patients, the presence, prevalence, severity, and morphological characteristics of anemia, trying to define, when possible, the underlying pathogenetic mechanisms, paying particular attention to the characteristics of menstrual cycles, the iron, folate and vitamin B12 metabolism, any chronic inflammatory state, and thyroid hormones. It will be also recorded, in a subgroup of the selected CD patients, any therapeutic responses (i.e., improvement/regression) of anemia after at least one year of GFD.

ELIGIBILITY:
Inclusion Criteria:

CD will be diagnosed according to the current guidelines. In details, the following standard criteria will be adopted to diagnose CD ("4 out of 5" rule):

* gluten/wheat-dependent symptoms, both intestinal and extraintestinal
* positivity of anti-deamidated gluten peptides (DPG) IgA and IgG antibodies, anti-transglutainase (tTG) IgA and IgG antibodies, and endomysium antibodies (EMA)
* presence of crypt hyperplasia and duodenal villous atrophy on duodenal biopsy
* presence of HLA haplotypes DQ2 and/or DQ8
* resolution of symptoms with a rigorous GFD

Additional inclusion criteria, both for the retrospective and prospective part of the study, will be:

* age >18 and <65 years
* complete clinical records
* clinical and laboratory follow-up of at least one year from diagnosis -

Exclusion Criteria:

* age <18 and >65 years
* incomplete medical records
* lack of clinical and laboratory follow-up of at least one year from diagnosis
* pregnancy
* alcohol and/or drug abuse
* diagnosis of IBD or other gastrointestinal organic disease

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will enroll CD patients.
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Presence, severity and morphologic characteristic of anemia | At baseline (=before diagnosis, on a gluten-containing diet) and at follow-up (=after at least one year of GFD)
  Blood count to evaluate red cell count and morphology

SECONDARY OUTCOMES:
Pathogenic mechanisms of anemia | At baseline (=before diagnosis, on a gluten-containing diet) and at follow-up (=after at least one year of GFD)
  Evaluation of inadequate production or loss of erythrocytes a a result of bleeding or hemolysis

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, MD, Study Director — University of Palermo
Locations (3):
- Italy (3):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Internal Medicine Division of the "Cervello-Villa Sofia" Hospital, Palermo, PA
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Montoro-Huguet MA, Santolaria-Piedrafita S, Canamares-Orbis P, Garcia-Erce JA. Iron Deficiency in Celiac Disease: Prevalence, Health Impact, and Clinical Management. Nutrients. 2021 Sep 28;13(10):3437. doi: 10.3390/nu13103437. PMID 34684433
- [Result] Martin-Masot R, Nestares MT, Diaz-Castro J, Lopez-Aliaga I, Alferez MJM, Moreno-Fernandez J, Maldonado J. Multifactorial Etiology of Anemia in Celiac Disease and Effect of Gluten-Free Diet: A Comprehensive Review. Nutrients. 2019 Oct 23;11(11):2557. doi: 10.3390/nu11112557. PMID 31652803
- [Result] Elli L, Norsa L, Zullo A, Carroccio A, Girelli C, Oliva S, Romano C, Leandro G, Bellini M, Marmo R, Soncini M, Monica F, De Francesco V, Paulon E, Cappellini MD, Motta I, Ferretti F, Orlando S, Mansueto P, Buscarini E, Manfredi G, Agostoni C, Tomba C, Cannizzaro R. Diagnosis of chronic anaemia in gastrointestinal disorders: A guideline by the Italian Association of Hospital Gastroenterologists and Endoscopists (AIGO) and the Italian Society of Paediatric Gastroenterology Hepatology and Nutrition (SIGENP). Dig Liver Dis. 2019 Apr;51(4):471-483. doi: 10.1016/j.dld.2019.01.022. Epub 2019 Feb 11. PMID 30850345
- [Result] Stefanelli G, Viscido A, Longo S, Magistroni M, Latella G. Persistent Iron Deficiency Anemia in Patients with Celiac Disease Despite a Gluten-Free Diet. Nutrients. 2020 Jul 22;12(8):2176. doi: 10.3390/nu12082176. PMID 32708019